CLINICAL TRIAL: NCT06016855
Title: Surgical Debulking Prior to Peptide Receptor Radionuclide Therapy (PRRT) in Patients With Well Differentiated Gastroenteropancreatic Neuroendocrine Tumors
Brief Title: Surgical Debulking Prior to Peptide Receptor Radionuclide Therapy in Well Differentiated Gastroenteropancreatic Neuroendocrine Tumors
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Principal Investigator, Kamran Idrees, Associate Professor of Surgery, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICCGI2283; NCI-2023-05914 (Registry Identifier: NCI, Clinical Trials Reporting Program)
Record Dates: First submitted 2023-08-23; First posted 2023-08-30 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Digestive System Neuroendocrine Tumor G1; Digestive System Neuroendocrine Tumor G2; Metastatic Digestive System Neuroendocrine Neoplasm; Metastatic Malignant Neoplasm in the Liver; Pancreatic Neuroendocrine Tumor G1; Pancreatic Neuroendocrine Tumor G2
MeSH Terms: interventions — lutetium Lu 177 dotatate; Magnetic Resonance Spectroscopy; 64Cu-DOTATATE

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (surgical debulking, 177Lu dotatate) (Experimental): Patients undergo surgical debulking on day 0 and receive 177Lu dotatate IV over 30 to 40 minutes on day 1 of each cycle. Treatment repeats every 56 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan or MRI throughout the trial, and undergo dotatate PET/CT during screening and on study.
  Interventions: Procedure: Tumor Debulking; Drug: Lutetium Lu 177 Dotatate; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Copper Cu 64 Dotatate; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Tumor Debulking — Undergo surgical debulking
Drug: Lutetium Lu 177 Dotatate — Given by IV
Procedure: Computed Tomography — Undergo Computed Tomography
Procedure: Magnetic Resonance Imaging — Undergo Magnetic Resonance Imaging
Drug: Copper Cu 64 Dotatate — Given by IV
Procedure: Positron Emission Tomography — Undergo Positron Emission Tomography

SUMMARY:
This phase IV trial evaluates how well giving standard of care (SOC) peptide receptor radionuclide therapy (PRRT) after SOC surgical removal of as much tumor as possible (debulking surgery) works in treating patients with grade 1 or 2, somatostatin receptor (SSTR) positive, gastroenteropancreatic neuroendocrine tumors (GEP-NETs) that have spread from where they first started (primary site) to the liver (hepatic metastasis). Lutetium Lu 177 dotatate is a radioactive drug that uses targeted radiation to kill tumor cells. Lutetium Lu 177 dotatate includes a radioactive form (an isotope) of the element called lutetium. This radioactive isotope (Lu-177) is attached to a molecule called dotatate. On the surface of GEP-NET tumor cells, a receptor called a somatostatin receptor binds to dotatate. When this binding occurs, the lutetium Lu 177 dotatate drug then enters somatostatin receptor-positive tumor cells, and radiation emitted by Lu-177 helps kill the cells. Giving lutetium Lu 177 dotatate after surgical debulking may better treat patients with grade 1/2 GEP-NETs

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To measure objective response rate of a combination standard of care treatment in gastroenteropancreatic neuroendocrine tumors by initiating lutetium Lu 177 dotatate within 90 days of surgical debulking.

II. To assess the radiomic profile including somatostatin receptor standardized uptake values (SSTR SUV) of large and non-large tumors in study patients)

III: To assess the safety and tolerability of peptide receptor radionuclide therapy (PRRT) post-surgical debulking in patients on study.

IV. To assess the tumor genomic profile of large, resected tumors from patients and assess for signatures of radioresistance.

OUTLINE:

Patients undergo surgical debulking on day 0 and receive lutetium Lu 177 dotatate (177Lu dotatate) intravenously (IV) over 30 to 40 minutes on day 1 of each cycle. Treatment repeats every 56 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) scan or magnetic resonance imaging (MRI) throughout the trial, and undergo copper Cu 64 dotatate positron emission tomography/CT (dotatate PET/CT) during screening and on study.

After completion of study treatment, patients are followed up at 30-37 days after last dose and then every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent
* Male or female >= 18 years of age on the day of signing informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Histologically confirmed well-differentiated gastrointestinal or pancreatic neuroendocrine tumor that is grade 1 or grade 2 (Ki-67 =< 20%)
* Somatostatin receptor avidity of known or suspected neuroendocrine tumor (NET) lesion(s) assessed by a baseline copper-64 dotatate PET/CT scan performed within 6 months (180 days) prior to surgical debulking on study day 0. The somatostatin receptor avidity of the majority of suspected NET lesion(s) must be >= normal liver uptake
* Patient must have hepatic metastasis or hepatic metastases. Provided required hepatic metastatic disease is present, patient can also have any other site or sites of metastatic disease
* White blood cell count (WBC) >= 2000/uL (resulted =< 90 days prior to surgical debulking on day 0 of participation in this study)
* Platelets >= 75,000/uL (resulted =< 90 days prior to surgical debulking on day 0 of participation in this study)
* Hemoglobin >= 8.0 g/dL (resulted =< 90 days prior to surgical debulking on day 0 of participation in this study)
* Creatinine clearance (CrCl) >= 30 mL/minute (as calculated by the Cockcroft-Gault Formula with estimated creatinine clearance rate [eCCR] >= 30 mL/min required for eligibility inclusion; or calculated/measured by an alternative established institutional standard consistently applied across participants at the site) (resulted =< 90 days prior to surgical debulking on day 0 of participation in this study)
* Total bilirubin =< 3.0 times institutional upper limit of normal (ULN) (resulted =< 90 days prior to surgical debulking on day 0 of participation in this study)
* Serum albumin >= 3.0 g/dL unless the prothrombin time is within normal range (resulted =< 90 days prior to surgical debulking on day 0 of participation in this study)
* Women must not be breastfeeding and further agree to not breastfeed during treatment with lutetium Lu 177 dotatate; and for at least 2.5 months after patient's final dose of lutetium Lu 177 dotatate
* A woman of childbearing potential (WOCBP) - must have a negative serum or urine pregnancy test resulted within 28 days prior to initiation of first dose of lutetium Lu 177 dotatate on cycle 1, day 1; and must agree to follow instructions for using acceptable contraception from the time of signing consent, and until 7 months after her final dose of lutetium Lu 177 dotatate
* A man able to father children who is sexually active with a WOCBP must agree to follow instructions for using acceptable contraception, from the time of signing consent, and until 4 months after his final dose of lutetium Lu 177 dotatate

Exclusion Criteria:

* Patient has any tumor > 3 cm deemed to be inoperable
* Patient has disease which is considered to be completely surgically resectable
* Patient has grade 3 neuroendocrine neoplasm (well-differentiated or poorly-differentiated tumor)
* Prior receipt of peptide receptor radionuclide therapy (PRRT)
* Patient possesses untreated or growing brain metastases (growth within 90 days prior to surgical debulking on day 0 of participation in this study)
* Unstable angina, congestive heart failure with New York Heart Association (NYHA) functional classification III or IV, or uncontrolled symptomatic cardiac arrythmia
* Any other significant medical, psychiatric, or surgical condition, currently uncontrolled by treatment, which in the judgment of the patient's study physician may reasonably be expected to interfere with patient's completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2027-05-28 (Estimated); Study Completion 2028-05-28 (Estimated)

PRIMARY OUTCOMES:
Somatostatin receptor standardized uptake values (SSTR SUV) | Up to 2 years
  SSTR SUV (not limited to but including measures such as SSTR SUV max, SSTR SUV mean) will be estimated for the patients undergoing post-operative research dotatate scans and compared to values from peptide receptor radionuclide therapy (PRRT) eligibility-conferring dotatate scans in these same patients. These quantitative analytics will be performed by central review. Changes in SSTR SUV values will be analyzed with summary statistics.
Progression-free survival | From the start of PRRT to the date the patient progresses radiographically or succumbs to the disease, assessed up to 2 years
  Will be estimated by the Kaplan-Meier method.
Overall response rate | Up to 2 years
  Will be estimated by measuring the number of patients who achieve a complete response or partial response by Response Evaluation Criteria in Solid Tumors (RECIST 1.1) criteria on restaging computed tomography or magnetic resonance imaging scans =< 6 months from PRRT completion, from the total number of patients who received the study treatment and possessed measurable disease post-surgical debulking. The number of patients who possessed measurable disease which did not meet RECIST 1.1 eligibility criteria post-surgical debulking will also be recorded.
Overall survival | From the start of PRRT to the date the patient progresses radiographically or succumbs to the disease, assessed up to 2 years
  Will be estimated by the Kaplan-Meier method.
Incidence of adverse events | Up to 2 years
  Toxicity will be estimated by documenting the grade 3/4 adverse events, according to Common Terminology Criteria for Adverse Events version 5.0, experienced by study patients.
Gene mutations | Up to 2 years
  Mutations in genes associated with radioresistance (defined from other malignancies) and other mutations in large resected neuroendocrine tumors will be recorded. Mutations will be described descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Kamran Idrees, MD, Principal Investigator — Vanderbilt University/Ingram Cancer Center
Locations (1):
- Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] von Hessert-Vaudoncourt C, Maasberg S, Begum N, Rinke A, Poppel T, Sipos B, Grohe C, Fottner C, Stintzing S, Grabowski P; German NET Registry. Clinical characteristics and treatment patterns of patients with gastroenteropancreatic neuroendocrine neoplasia in Germany receiving peptide receptor radionuclide therapy: A real-world data registry-based study. Medicine (Baltimore). 2025 Mar 14;104(11):e41853. doi: 10.1097/MD.0000000000041853. PMID 40101049

DOCUMENTS (1):
  • Informed Consent Form (2023-07-14): https://cdn.clinicaltrials.gov/large-docs/55/NCT06016855/ICF_000.pdf